CLINICAL TRIAL: NCT00907478
Title: A Prospective, Phase IV, Open-Label, Multi-Center Study Evaluating Changes in Bone Marrow Morphology in Adult Subjects Receiving Romiplostim for the Treatment of Thrombocytopenia Associated With Immune (Idiopathic) Thrombocytopenia Purpura (ITP)
Brief Title: Study on Bone Marrow Morphology in Adults Receiving Romiplostim for Treatment of Thrombocytopenia Associated With Immune Thrombocytopenia Purpura (ITP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080009
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Thrombocytopenia; Idiopathic Thrombocytopenic Purpura
Keywords: Idiopathic Thrombocytopenic Purpura; Idiopathic Thrombocytopenia Purpura; Immune Thrombocytopenic Purpura; Immune Thrombocytopenia; ITP
MeSH Terms: conditions — Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romiplostim (Experimental): Participants received romiplostim administered weekly by subcutaneous injection for up to 3 years.
  The starting dose of romiplostim was 1 μg/kg; weekly dose increases continued in increments of 1 μg/kg/week to a maximum dose of 10 μg/kg in an attempt to reach a target platelet count of ≥ 50 x 10^9/L.
  Interventions: Biological: romiplostim

INTERVENTIONS:
Biological: romiplostim — Romiplostim administered by subcutaneous injection
  Other Names: Nplate®

SUMMARY:
The purpose of this study is to evaluate changes in bone marrow morphology (structure) after long-term exposure to romiplostim.

DETAILED DESCRIPTION:
Participants diagnosed with ITP according to the American Society of Hematology (ASH) Guidelines were sequentially enrolled into the following groups:

* Bone marrow biopsy at Baseline and Year 1
* Bone marrow biopsy at Baseline and Year 2
* Bone marrow biopsy at Baseline and Year 3.

All participants received romiplostim for 3 years, unless withdrawn from the study early. Participants returned for one visit for End of Study (EOS) procedures 4 weeks after romiplostim discontinuation, or, for participants who were withdrawn from the study due to the presence of collagen fibrosis, or had a change to grade 3 reticulin, at 12 weeks after discontinuation of romiplostim.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ITP according to American Society of Hematology (ASH) guidelines
* Subject must have had a bone marrow biopsy within one year prior to planned first dose of romiplostim (with available bone marrow tissue block or unstained histological slides to send to a central laboratory for interpretation) or must consent to a pre-treatment bone marrow biopsy within 3 weeks prior to planned first dose of romiplostim. Central laboratory interpretation is required prior to first dose of romiplostim
* Subject must agree to a scheduled bone marrow biopsy at Year 1, Year 2, or Year 3 following romiplostim treatment and any unscheduled biopsies if clinically indicated
* Subject ≥18 years of age
* Baseline bone marrow reticulin grade of 0, 1, 2, or 3 according to the modified Bauermeister grading scheme as assessed by central laboratory interpretation
* Platelet count < 50 x 10^9/L
* Must have received at least 1 prior ITP therapy (examples of ITP therapy include corticosteroids, intravenous immunoglobulin [IVIG], splenectomy)
* Subject (or legally-acceptable representative) is willing and able to provide written informed consent

Exclusion Criteria:

* Baseline bone marrow biopsy positive for collagen fibrosis
* Any known history of or currently active bone marrow stem cell disorder, hematological malignancy, myeloproliferative disorder, myelodysplastic syndrome
* Any current active malignancy
* Any prior exposure to cytostatic chemotherapy or radiotherapy for malignancy
* Subject has undergone pacemaker placement, cardiac ablation of arrhythmia, and/or any current treatment with Vaughan Williams Class IA - IC and Class III agents (Vaughan Williams, 1970)
* Subject has participated in any study evaluating pegylated recombinant human megakaryocyte growth and development factor (PEG-rHuMGDF), recombinant human thrombopoietin (rHuTPO), or thrombopoietin receptor agonists (ie romiplostim or eltrombopag)
* Subject has a known hypersensitivity to any recombinant E coli-derived product
* Subject is currently enrolled in or has not yet completed (at least 4 weeks since ending) other investigational device or drug trial(s) or subject is receiving other investigational agent(s)
* Other investigational procedures are excluded
* Subject of child-bearing potential is evidently pregnant (eg positive pregnancy test) or is breast feeding
* Subject is not using adequate contraceptive precautions
* Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and does not have a legally acceptable representative and/or is unable to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2009-08-11 (Actual); Primary Completion 2014-01-09 (Actual); Study Completion 2014-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Janssens A, Rodeghiero F, Anderson D, Chong BH, Boda Z, Pabinger I, Cervinek L, Terrell DR, Wang X, Franklin J. Changes in bone marrow morphology in adults receiving romiplostim for the treatment of thrombocytopenia associated with primary immune thrombocytopenia. Ann Hematol. 2016 Jun;95(7):1077-87. doi: 10.1007/s00277-016-2682-2. Epub 2016 Apr 30. PMID 27130310
- [Background] Cines DB, Wasser J, Rodeghiero F, Chong BH, Steurer M, Provan D, Lyons R, Garcia-Chavez J, Carpenter N, Wang X, Eisen M. Safety and efficacy of romiplostim in splenectomized and nonsplenectomized patients with primary immune thrombocytopenia. Haematologica. 2017 Aug;102(8):1342-1351. doi: 10.3324/haematol.2016.161968. Epub 2017 Apr 14. PMID 28411254
- [Background] Kuter DJ, Newland A, Chong BH, Rodeghiero F, Romero MT, Pabinger I, Chen Y, Wang K, Mehta B, Eisen M. Romiplostim in adult patients with newly diagnosed or persistent immune thrombocytopenia (ITP) for up to 1 year and in those with chronic ITP for more than 1 year: a subgroup analysis of integrated data from completed romiplostim studies. Br J Haematol. 2019 May;185(3):503-513. doi: 10.1111/bjh.15803. Epub 2019 Feb 21. PMID 30793285
- [Background] Kuter DJ, Arnold DM, Rodeghiero F, Janssens A, Selleslag D, Bird R, Newland A, Mayer J, Wang K, Olie R. Safety and efficacy of self-administered romiplostim in patients with immune thrombocytopenia: Results of an integrated database of five clinical trials. Am J Hematol. 2020 Jun;95(6):643-651. doi: 10.1002/ajh.25776. Epub 2020 Mar 21. PMID 32129511
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were adults diagnosed with immune (idiopathic) thrombocytopenic purpura (ITP) with a platelet count < 50 x 10^9/L. The first patient enrolled 11 August 2009 and the last patient was enrolled 11 November 2010. Participants were enrolled at 60 study centers in Australia, Europe, and North America.
Pre-assignment Details: 204 patients were screened, 35 were considered screen failures. Participants were enrolled sequentially into the following cohorts: • Bone marrow biopsy at Baseline and Year 1 • Bone marrow biopsy at Baseline and Year 2 • Bone marrow biopsy at Baseline and Year 3.
Groups:
- Cohort 1: Participants received once weekly romiplostim for 3 years and had a bone marrow biopsy at Baseline and Year 1.
- Cohort 2: Participants received once weekly romiplostim for 3 years and had a bone marrow biopsy at Baseline and Year 2.
- Cohort 3: Participants received once weekly romiplostim for 3 years and had a bone marrow biopsy at Baseline and Year 3.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 50 | 50 | 69
Completed | 23 (Defined as participants who completed the full 3 years and completed the end of study visit.) | 33 (Defined as participants who completed the full 3 years and completed the end of study visit.) | 47 (Defined as participants who completed the full 3 years and completed the end of study visit.)
Not Completed | 27 | 17 | 22
Not completed — Ineligibility determined | 0 | 0 | 1
Not completed — Noncompliance | 0 | 0 | 1
Not completed — Adverse Event | 3 | 1 | 2
Not completed — Withdrawal by Subject | 8 | 9 | 6
Not completed — Requirement for alternative therapy | 1 | 2 | 3
Not completed — Physician Decision | 2 | 0 | 3
Not completed — Death | 4 | 2 | 1
Not completed — Protocol-specified criteria | 5 | 2 | 3
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 50 | 50 | 69 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (17.1) | 48.6 (16.5) | 46.6 (16.3) | 49.8 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 38 | 49 | 114
  Male | 23 | 12 | 20 | 55
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 48 | 47 | 59 | 154
  Black or African American | 0 | 0 | 1 | 1
  Hispanic or Latino | 1 | 3 | 7 | 11
  Asian | 1 | 0 | 1 | 2
  Other | 0 | 0 | 1 | 1
Time Since ITP Diagnosis [Mean (Standard Deviation); unit: years] | 9.94 (10.29) | 10.50 (11.87) | 5.36 (6.41) | 8.24 (9.72)
Number of Prior ITP Therapies [Number; unit: participants]
  0 | 0 | 0 | 0 | 0
  1 | 16 | 16 | 29 | 61
  2 | 11 | 15 | 20 | 46
  3 | 8 | 9 | 10 | 27
  ≥ 4 | 15 | 10 | 10 | 35
Had Splenectomy [Number; unit: participants]
  No | 28 | 35 | 46 | 109
  Yes | 22 | 15 | 23 | 60
Any Prior History of Bone Marrow Abnormalities [Number; unit: participants]
  No | 48 | 47 | 64 | 159
  Yes | 2 | 3 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Collagen Fibrosis
Description: The percentage of participants who developed collagen fibrosis as evidenced by trichrome staining. Bone marrow biopsy samples were assessed using the modified Bauermeister grading scale by a central laboratory.
Time Frame: At Years 1, 2 or 3 after initial exposure of romiplostim
Population: Participants who had evaluable trichrome stain results
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 35 | 39 | 58
percentage of participants | 0.0 [0.0 to 10.0] | 0.0 [0.0 to 9.0] | 3.4 [0.4 to 11.9]

2. Secondary Outcome: Number of Participants With Collagen Fibrosis 12 Weeks After Romiplostim Discontinuation in Participants Who Developed Collagen Fibrosis at Years 1, 2, or 3
Description: The number of participants with collagen fibrosis as evidenced by trichrome staining 12 weeks after romiplostim discontinuation in participants who developed collagen fibrosis at Years 1, 2, or 3 after initial exposure of romiplostim, assessed by the central laboratory using the modified Bauermeister grading scale.
Time Frame: 12 weeks after romiplostim discontinuation
Population: Participants with collagen fibrosis at Year 1, 2 or 3 and with available trichome staining results 12 weeks after study drug discontinuation. One participant with collagen fibrosis refused the follow-up bone marrow biopsy.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 1
participants |  |  | 0

3. Secondary Outcome: Percentage of Participants Who Developed an Increased Modified Bauermeister Grade
Description: Increased modified Bauermeister grade refers to an increase by ≥ 2 severity grades or an increase to grade 4 (ie, grade 0 to 2-4, grade 1 to 3-4, grade 2 to 4, or grade 3 to 4 over baseline). The modified Bauermeister scale provides a means of assessing the development of increased reticulin and collagen in bone marrow according to the following: Grade 0: No reticulin fibers demonstrable; Grade 1: Occasional fine individual fibers and foci of a fine fiber network; Grade 2: Fine fiber network throughout most of the section; no coarse fibers; Grade 3: Diffuse fiber network with scattered thick coarse fibers but no mature collagen (negative to trichrome staining); Grade 4: Diffuse, often course fiber network with areas of collagenization (positive trichrome staining).
Time Frame: At Year 1, Year 2, or Year 3 post romiplostim exposure
Population: Participants who had evaluable reticulin silver stain results
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 34 | 39 | 58
percentage of participants | 0.0 [0.0 to 10.3] | 5.1 [0.6 to 17.3] | 12.1 [5.0 to 23.3]

4. Secondary Outcome: Percentage of Participants With Clinically Relevant Changes in Total Cardiac Output Corrected (QTc) Intervals
Description: A clinically relevant change in QTc (Fridericia) interval is defined as an absolute QTc interval >500 ms or a QTc Interval increase from Baseline >60 ms post romiplostim exposure. 12-lead electrocardiograms (ECG) were performed in triplicate at Baseline, Week 3 and Week 12; the average of of the 3 values at each assessment was used.
Time Frame: Baseline, Week 3 and Week 12
Population: All participants who received at least one dose of romiplostim.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 50 | 50 | 69
percentage of participants | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 5.2]

5. Secondary Outcome: Number of Participants With Improvement of Reticulin to a Grade of ≤ 2 for Participants Who Developed Grade 3 Reticulin
Description: The number of participants who had any improvement of reticulin to a grade of ≤ 2 for participants who developed grade 3 reticulin after initial exposure to romiplostim as measured by the modified Bauermeister grading scale. The modified Bauermeister scale provides a means of assessing the development of increased reticulin and collagen in bone marrow according to the following: Grade 0: No reticulin fibers demonstrable; Grade 1: Occasional fine individual fibers and foci of a fine fiber network; Grade 2: Fine fiber network throughout most of the section; no coarse fibers; Grade 3: Diffuse fiber network with scattered thick coarse fibers but no mature collagen (negative to trichrome staining); Grade 4: Diffuse, often course fiber network with areas of collagenization (positive trichrome staining).
Time Frame: 12 weeks after romiplostim discontinuation
Population: Participants with Grade 3 reticulin at Year 1, 2 or 3 and who had a follow-up bone marrow biopsy 12 weeks after romiplostim discontinuation. Two participants with grade 3 reticulin did not have a bone marrow biopsy performed 12 weeks after romiploastim discontinuation.
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 0 | 0 | 3
participants |  |  | 3

6. Secondary Outcome: Percentage of Participants With CTCAE Grade ≥ 2 Shift in Anemia or Neutropenia
Description: Anemia was identified by laboratory values with hemoglobin < the lower limit of normal (LLN) or the Medical Dictionary for Regulatory Activities (MedDRA) terms prespecified by the sponsor. Neutropenia was identified by laboratory values with absolute neutrophil count <1.8x10^9/L or the MedDRA terms pre-specified by the sponsor. Severity was assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, based on the following: Grade 1: Mild AE; Grade 2: Moderate AE; Grade 3: Severe AE; Grade 4: Life-threatening or disabling AE; Grade 5: Death related to AE.
Time Frame: From the first dose of study drug until 4 weeks after treatment discontinuation or 12 weeks after treatment discontinuation for patients who developed collagen fibrosis or a change to grade 3 reticulin; the overall median treatment duration was 154 weeks.
Population: All participants who received at least one dose of romiplostim
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 50 | 50 | 69
percentage of participants
  CTCAE grade ≥2 shift in anemia | 6.0 [1.3 to 16.5] | 4.0 [0.5 to 13.7] | 8.7 [3.3 to 18.0]
  CTCAE grade ≥2 shift in neutropenia | 8.0 [2.2 to 19.2] | 6.0 [1.3 to 16.5] | 13.0 [6.1 to 23.3]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant that did not necessarily have a causal relationship with this treatment, or any such occurrence or worsening of a pre-existing medical condition from the first dose of investigational product through the last study visit. A serious adverse event is defined as an AE that is fatal or life threatening, requires or prolongs hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or other significant medical hazard. The relationship of each AE to the study drug was assessed by the investigator. The severity of each AE was graded using using CTCAE 3.0; For any AEs not listed in CTCAE, the Amgen Standard Severity Scoring System was used: 1: Mild- Aware of sign or symptom, but easily tolerated; 2 Moderate- Discomfort enough to cause interference with usual activity; 3: Severe- Incapacitating with inability to work or do usual activity; 4: Life-threatening; 5: Fatal.
Time Frame: as for outcome 6
Population: All participants who received at least one dose of romiplostim
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 50 | 50 | 69
participants
  All adverse events | 46 | 45 | 67
  Grade ≥ 2 | 39 | 39 | 59
  Grade ≥ 3 | 25 | 21 | 38
  Grade ≥ 4 | 13 | 8 | 16
  Serious adverse events | 16 | 12 | 28
  Leading to discontinuation of study drug | 6 | 5 | 4
  Leading to discontinuation from study | 6 | 2 | 3
  Fatal adverse events | 4 | 2 | 1
  Treatment-related adverse events | 14 | 22 | 24
  Treatment-related grade ≥ 2 | 8 | 14 | 10
  Treatment-related grade ≥ 3 | 2 | 7 | 3
  Treatment-related grade ≥ 4 | 0 | 1 | 0
  Treatment-related serious adverse events | 1 | 2 | 3
  Treatment-related -> discontinuation of study drug | 1 | 1 | 2
  Treatment-related -> discontinuation from study | 1 | 0 | 2
  Treatment-related fatal adverse events | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Who Developed Antibodies or Neutralizing Antibodies to Romiplostim or to Endogenous Thrombopoietin
Description: Two validated assays were used to test for antibodies to romiplostim, the thrombopoietin-mimetic peptide component of romiplostim (TMP) and to endogenous thrombopoietin (TPO). The first was an immunoassay to confirm the presence of antibodies. The second was a cell-based bioassay to detect neutralizing or inhibitory effects in vitro. If a sample was positive in both assays, a participant was defined as positive for neutralizing antibodies.
  Persistent antibodies were those positive at the last timepoint tested and transient are defined as positive post-dose but negative at the last time point tested.
Time Frame: Every 24 weeks and at the end of study visit (4 weeks or 12 weeks after study drug discontinuation).
Population: All participants who received at least one dose of romiplostim.
Measure: Number; unit: participants
Groups:
- Romiplostim: Participants received once weekly romiplostim for 3 years.
Arm/Group | Romiplostim
Number analyzed (Participants) | 169
participants
  Antibodies to romiplostim | 7
  Persistent antibodies to romiplostim | 4
  Transient antibodies to romiplostim | 3
  Antibodies to TMP | 4
  Persistent antibodies to TMP | 1
  Transient antibodies to TMP | 3
  Antibodies to TPO | 6
  Persistent antibodies to TPO | 2
  Transient antibodies to TPO | 4
  Neutralizing antibodies to romiplostim | 1
  Neutralizing antibodies to TPO | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 4 weeks after treatment discontinuation or 12 weeks after treatment discontinuation for patients who developed collagen fibrosis or a change to grade 3 reticulin; the overall median treatment duration was 154 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Cohort 2: Year 1 Participants received once weekly romiplostim for 3 years and had a bone marrow biopsy at Baseline and Year 2.
- Cohort 3: Year 1 Participants received once weekly romiplostim for 3 years and had a bone marrow biopsy at Baseline and Year 3.
- Overall: Participants received once weekly romiplostim for 3 years.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Overall
Serious Adverse Events (participants affected / at risk) | 16/50 | 12/50 | 28/69 | 56/169
Other Adverse Events (participants affected / at risk) | 45/50 | 43/50 | 66/69 | 154/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=50) | Cohort 2 (N=50) | Cohort 3 (N=69) | Overall (N=169)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 3
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Haemorrhagic Diathesis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 1 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 4 | 6
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 2 | 2
Atrial Flutter (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac Disorder (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 1
Conjunctival Haemorrhage (Eye disorders) | 0 | 0 | 1 | 1
Glaucoma (Eye disorders) | 1 | 0 | 0 | 1
Hyphaema (Eye disorders) | 1 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Acute Abdomen (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gingival Disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 2 | 2
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Abscess Jaw (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 1
Fungal Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Lobar Pneumonia (Infections and infestations) | 1 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 2
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 0 | 3
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Clostridium Test Positive (Investigations) | 1 | 0 | 0 | 1
Weight Decreased (Investigations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 2 | 0 | 0 | 2
Complicated Migraine (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 2
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 1 | 1
Sensory Disturbance (Nervous system disorders) | 0 | 0 | 1 | 1
Spinal Claudication (Nervous system disorders) | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Completed Suicide (Psychiatric disorders) | 0 | 1 | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Calculus Urethral (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 1 | 2
Adenomyosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Lichenoid Keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Knee Operation (Surgical and medical procedures) | 0 | 0 | 1 | 1
Tooth Extraction (Surgical and medical procedures) | 1 | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 2 | 2
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Peripheral Embolism (Vascular disorders) | 0 | 0 | 1 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 0 | 1 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=50) | Cohort 2 (N=50) | Cohort 3 (N=69) | Overall (N=169)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 4 | 8
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 8 | 6 | 8 | 22
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 4 | 7
Neutrophilia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 3 | 6 | 17
Palpitations (Cardiac disorders) | 1 | 1 | 4 | 6
Tachycardia (Cardiac disorders) | 3 | 0 | 1 | 4
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 5 | 7
Cataract (Eye disorders) | 3 | 2 | 2 | 7
Abdominal Pain (Gastrointestinal disorders) | 2 | 2 | 8 | 12
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 4 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 3 | 5 | 10
Constipation (Gastrointestinal disorders) | 3 | 3 | 5 | 11
Diarrhoea (Gastrointestinal disorders) | 7 | 7 | 18 | 32
Gingival Bleeding (Gastrointestinal disorders) | 3 | 5 | 13 | 21
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 4 | 5
Mouth Haemorrhage (Gastrointestinal disorders) | 6 | 5 | 2 | 13
Nausea (Gastrointestinal disorders) | 6 | 7 | 11 | 24
Vomiting (Gastrointestinal disorders) | 5 | 6 | 8 | 19
Chest Pain (General disorders) | 1 | 0 | 8 | 9
Fatigue (General disorders) | 6 | 8 | 7 | 21
Influenza Like Illness (General disorders) | 0 | 3 | 3 | 6
Local Swelling (General disorders) | 5 | 5 | 3 | 13
Malaise (General disorders) | 0 | 3 | 1 | 4
Oedema Peripheral (General disorders) | 4 | 3 | 4 | 11
Pain (General disorders) | 0 | 2 | 5 | 7
Pyrexia (General disorders) | 6 | 4 | 10 | 20
Bronchitis (Infections and infestations) | 3 | 9 | 12 | 24
Influenza (Infections and infestations) | 1 | 7 | 8 | 16
Nasopharyngitis (Infections and infestations) | 6 | 21 | 14 | 41
Pharyngitis (Infections and infestations) | 1 | 4 | 6 | 11
Respiratory Tract Infection (Infections and infestations) | 2 | 3 | 2 | 7
Sinusitis (Infections and infestations) | 3 | 5 | 7 | 15
Upper Respiratory Tract Infection (Infections and infestations) | 11 | 7 | 13 | 31
Urinary Tract Infection (Infections and infestations) | 4 | 6 | 6 | 16
Viral Infection (Infections and infestations) | 1 | 3 | 7 | 11
Contusion (Injury, poisoning and procedural complications) | 6 | 9 | 19 | 34
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 5 | 9
Laceration (Injury, poisoning and procedural complications) | 1 | 3 | 5 | 9
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 7 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3 | 2 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 10 | 19 | 37
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 11 | 24
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 9 | 12
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 7
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 5 | 8 | 17
Dizziness (Nervous system disorders) | 4 | 6 | 4 | 14
Headache (Nervous system disorders) | 12 | 14 | 25 | 51
Paraesthesia (Nervous system disorders) | 1 | 2 | 5 | 8
Insomnia (Psychiatric disorders) | 3 | 7 | 3 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 13 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 18 | 37
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 10 | 17
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 5 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 7
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 3 | 4 | 9
Petechiae (Skin and subcutaneous tissue disorders) | 9 | 11 | 14 | 34
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 6 | 8 | 15
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 7 | 14
Haematoma (Vascular disorders) | 2 | 3 | 10 | 15
Hypertension (Vascular disorders) | 0 | 4 | 5 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.